CLINICAL TRIAL: NCT00071058
Title: A Study of Combination Chemotherapy & Surgical Resection in the Tx of Adrenocortical Cancer: Mitotane & Continuous Infusion Doxorubicin, Vincristine & Etoposide w/the P-glycoprotein Antagonist, Tariquidar (XR9576), Before & After Surgical Resection
Brief Title: Surgery Plus Chemotherapy (Doxorubicin, Vincristine and Etoposide), Mitotane, and Tariquidar to Treat Adrenocortical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Antonio Fojo, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040011; 04-C-0011; NCT00073996 (obsolete NCT alias)
Record Dates: First submitted 2003-10-09; First posted 2003-10-10 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Adrenal Cortex Neoplasms
Keywords: P-glycoprotein Inhibition; Drug Resistance Reversal; Pharmacodynamics; Molecular Target; Endocrine Cancer; Adrenocortical Cancer; ACC; Adrenocortical Tumor
MeSH Terms: conditions — Adrenal Cortex Neoplasms; Endocrine Gland Neoplasms | interventions — tariquidar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery plus chemotherapy (Experimental): Surgical resection can be performed at the time of study entry, when patients have a mixed response, or if their tumors respond to chemotherapy.
  Surgical resection will be followed by chemotherapy with 2 grams oral dose daily of mitotane on cycle 1, day 1, 6 mg/m^2 continuous intravenous infusion doxorubicin over 96 hours days 1-4, 0.18 mg/m^2 continuous intravenous infusion vincristine over 96 hours days 1-4, and 36 mg/m^2 continuous intravenous infusion etoposide over 96 hours days 1-4, and 150 mg tariquidar through central venous catheter over 30 minutes on days 1 and 3.
  Interventions: Drug: XR9576 (Tariquidar)

INTERVENTIONS:
Drug: XR9576 (Tariquidar)
  Other Names: 150 mg tariquidar through central venous catheter over 30 minutes on days 1 and 3.

SUMMARY:
This study will examine the safety and effectiveness of treating adrenocortical cancer with combination chemotherapy using doxorubicin, vincristine, and etoposide in addition to the drugs mitotane and tariquidar and, when possible, surgery. Adrenocortical cancer cells have a large amount of a protein called P-glycoprotein that "pumps" anti-cancer drugs out of the cells, decreasing their effectiveness. Continuous infusions of doxorubicin, vincristine, and etoposide may improve chemotherapy results by blocking the P-glycoprotein pump, as may use of tariquidar, an experimental drug that is known to block the P-glycoprotein pump.

Patients 18 years of age and older with adrenocortical cancer that has recurred, spread, or cannot be treated surgically may be eligible for this study. Candidates will be screened with a medical history and physical examination; review of pathology slides; blood tests; electrocardiogram (EKG); imaging tests, including computed tomography (CT) of the chest, abdomen and pelvis; chest x-ray; and possibly a bone scan or other imaging tests needed to evaluate the cancer, urine studies, and an echocardiogram. Also, a biopsy (removal of a small sample of tumor tissue) may be required if a specimen is not available to confirm the cancer.

Participants will undergo the following tests and procedures:

* Tumor biopsy. Before starting chemotherapy, a small piece of tumor is removed to study the P-glycoprotein pump and to determine the tumor genetics.
* Blood draw. Blood is drawn before treatment begins to establish baseline levels for future blood tests.
* Central venous catheter placement. A specially trained physician places a plastic tube into a major vein in the chest. The tube is used to give the study drugs and other medications and to withdraw blood samples. It can stay in the body for months or be removed after each treatment is completed. The tube placement is done under a local anesthetic in the radiology department or operating room.
* Chemotherapy. Treatment cycles are 21 days. Doxorubicin, vincristine, and etoposide are given through the central venous catheter by an infusion pump continuously over 96 hours starting day 1 of each cycle. The dose of these drugs may be increased or decreased from cycle to cycle, based on side effects. Mitotane is given in pill form starting day 1 of cycle 1 and is taken every day throughout the entire study. The mitotane dose is gradually increased as long as the side effects are tolerable. Tariquidar is given through the central venous catheter as a 30-minute infusion on days 1 and 3 of every cycle. The tariquidar dose remains the same throughout the study. Treatment will continue for two cycles after all the cancer is gone, or until surgery is done to remove some or all of the remaining cancer, or, if surgery is not an option, until the cancer has grown to where it is defined as progressive disease.
* Nuclear scans. A nuclear scan is done before treatment begins and again on day 1 or day 3 of the first treatment cycle after administration of tariquidar to evaluate the P glycoprotein response to treatment.
* Computed tomography (CT) scans. These scans are done every two treatment cycles to follow disease progress.
* Surgery. Surgery to remove areas of cancer may be considered at any point during the study (including before beginning treatment), if it is deemed beneficial. Treatment with the study drugs will begin or resume after surgery. The length of treatment will depend on the response to treatment before the surgery and on whether there is any cancer remaining after the surgery.

DETAILED DESCRIPTION:
Adrenocortical cancer (ACC) is a rare tumor that is optimally treated with surgical resection. However, many patients present with unresectable disease and relapses are common after surgical resection creating a need for more effective systemic therapies. Several investigators have reported responses to a variety of chemotherapy agents, without a clear improvement in overall survival. A possible explanation for these disappointing results is the high levels of expression of P-glycoprotein (Pgp) seen in a majority of adrenocortical cancers. Pgp, a membrane protein that can function as a drug efflux pump lowering the intracellular concentrations of various drugs, has been implicated as a mechanism of drug resistance.

A prior National Cancer Institute (NCI) study (referred to as MAVE) tried to improve response rates by using a combined modality approach with chemotherapy and surgery. Prior in vitro studies had shown that mitotane inhibited Pgp and that continuous exposure to doxorubicin and vincristine was more effective at overcoming Pgp-mediated resistance than the same drugs given on an intermittent schedule. The MAVE study used daily oral mitotane with infusional doxorubicin, vincristine, and etoposide prior to tumor resection in patients with resectable or potentially resectable tumors. The results showed an overall response rate of 19% (including minor responses), and an overall median survival of 13.5 months. These results were similar to those reported with previous regimens in adrenocortical cancer (ACC). A possible explanation for the failure to achieve a higher response rate may be that mitotane was unable to inhibit Pgp. Although the serum levels of mitotane achieved in patients had been shown to block Pgp in vitro, inhibition of Pgp in patients was not accomplished, as documented by a validated surrogate assay using Pgp-expressing CD56+ cells and the Pgp substrate, rhodamine. Thus the question of whether Pgp inhibition would improve response rates remains unanswered.

This trial will attempt to answer the latter question by using an agent, tariquidar (XR9576), which has been proven to inhibit Pgp in humans with minimal toxicity alone or in combination with chemotherapy. Tariquidar will be used with the regimen from the prior MAVE study in an effort to improve response rates and overall survival in patients with ACC whose options at this time are limited.

ELIGIBILITY:
* INCLUSION CRITERIA:

Pathologic confirmation of adrenocortical cancer by the Laboratory of Pathology, NCI

Diagnosis of recurrent, metastatic, or primary unresectable adrenocortical carcinoma.

Measurable disease at presentation.

A life expectancy of at least 3 months and Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.

Age greater than or equal to 18 years.

Last dose of chemotherapy or experimental therapy more than 4 weeks (6 weeks in the case of nitrosourea) prior to enrollment date.

Last radiotherapy treatment 4 weeks prior to starting treatment with this protocol and there must be sites of measurable disease that did not receive radiation.

Prior mitotane therapy is allowed. Patients do not need to be off mitotane therapy prior to starting this protocol.

Organ and marrow function as defined below:

* Total bilirubin less than or equal to 1.5 times ULN (upper limit of normal), unless the patient meets the criteria for Gilbert's Syndrome,
* Aspartate aminotransferase (AST) less than or equal to 3 times ULN, Alanine aminotransferase (ALT) less than or equal to 3 times ULN
* Creatinine clearance greater than or equal to 40 ml/min (measured in a timed urine collection) or serum creatinine less than or equal to 1.6 mg/dl
* Absolute neutrophil count greater than or equal to 1000/mm^3,
* Platelet count greater than or equal to 100,000/mm^3

Ability to understand and sign an informed consent document.

Ability and willingness to follow the guidelines of the clinical protocol including visits to National Cancer Institute (NCI), Bethesda, Maryland for treatment and follow up visits.

The effects of chemotherapy on the developing human fetus are potentially harmful therefore women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier methods) during the study and for a period of 1 month after the last dose of chemotherapy.

EXCLUSION CRITERIA:

Patients with adrenocortical tumors potentially curable by surgical excision alone as determined by the Principal Investigator in discussions with the surgical consultants.

Uncontrolled illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, seizure disorder, or psychiatric illness that may limit compliance with study requirements. These illnesses may be exacerbated by chemotherapy.

Untreated brain metastases (or local treatment of brain metastases within the last 6 months) due to the poor prognosis of these patients and difficulty ascertaining the cause of neurologic toxicities.

Pregnancy due to the possible adverse effects on the developing fetus.

Lactating women who are breast-feeding due to the possibility of transmitting chemotherapy to the child.

The presence of a second malignancy, other than squamous cell carcinoma of the skin or in situ cervical cancer because it will complicate the primary objective of the study. Cancer survivors who have been free of disease for at least two years can be enrolled in this study.

Currently receiving treatment (which cannot be discontinued) with the following agents: diltiazem, nicardipine, phenothiazines, phenytoin, or verapamil because these are Pgp inhibitors and will interfere with the primary objective of the study.

Ejection fraction less than 40% as determined by multi-gated acquisition scan (MUGA), echocardiogram (Echo), or cardiac magnetic resonance imaging (MRI) in patients with a clinical history suggestive of systolic dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Fojo, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Cohn K, Gottesman L, Brennan M. Adrenocortical carcinoma. Surgery. 1986 Dec;100(6):1170-7. PMID 3787475
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_2004-C-0011.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surgery Plus Chemotherapy
Started | 50
Completed | 49
Not Completed | 1
Not completed — brain tumor-removed from study | 1

BASELINE CHARACTERISTICS:
Groups:
- Surgery Plus Chemothrapy: Surgical resection can be performed at the time of study entry, when patients have a mixed response, or if their tumors respond to chemotherapy.
  Surgical resection will be followed by chemotherapy with 2 grams oral dose daily of mitotane on cycle 1, day 1, 6 mg/m^2 continuous intravenous infusion doxorubicin over 96 hours days 1-4, 0.18 mg/m2 continuous intravenous infusion vincristine over 96 hours days 1-4, and 36 mg/m^2 continuous intravenous infusion etoposide over 96 hours days 1-4, and 150 mg tariquidar through central venous catheter over 30 minutes on days 1 and 3.
Arm/Group | Surgery Plus Chemothrapy
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 45.56 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Partial or Complete Response
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Complete response is defined as the disappearance of all signs and symptoms of tumor for a period of at least 4 weeks. Partial response is defined as at least a 30% decrease in the sum of the longest diameter of all measured lesions lasting for a period of 4 weeks.
Time Frame: Every 6 weeks for up to a year
Measure: Number; unit: Percentage of participants
Groups:
- Surgery Plus Chemotherapy: Surgical resection can be performed at the time of study entry, when patients have a mixed response, or if their tumors respond to chemotherapy.
  Surgical resection will be followed by chemotherapy with 2 grams oral dose daily of mitotane on cycle 1, day 1, 6 mg/m^2 continuous intravenous infusion doxorubicin over 96 hours days 1-4, 0.18 mg/m2 continuous intravenous infusion vincristine over 96 hours days 1-4, and 36 mg/m^2 continuous intravenous infusion etoposide over 96 hours days 1-4, and 150 mg tariquidar through central venous catheter over 30 minutes on days 1 and 3.
Arm/Group | Surgery Plus Chemotherapy
Number analyzed (Participants) | 49
Percentage of participants
  Complete Response | 4
  Partial Response | 6

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 60 months, 19 days
Measure: Number; unit: Participants
Arm/Group | Surgery Plus Chemotherapy
Number analyzed (Participants) | 49
Participants | 49

ADVERSE EVENTS:
Arm/Group | Surgery Plus Chemothrapy
Serious Adverse Events (participants affected / at risk) | 13/50
Other Adverse Events (participants affected / at risk) | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery Plus Chemothrapy (N=50)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3 (3)
Cardiac left ventricular function (Cardiac disorders) | 1 (1)
Cardiac-ischemia/infarction (Cardiac disorders) | 1 (2)
Thrombosis/embolism (Cardiac disorders) | 2 (2)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 5 (5)
Rigors/chills (General disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 1 (1)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 1 (1)
Ileus (or neuroconstipation) (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 3 (3)
Febrile Neutropenia (Infections and infestations) | 2 (2) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Infection (Infections and infestations) | 1 (1) — (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e9/L)
Infection without neutropenia (Infections and infestations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Abdominal pain or cramping (Gastrointestinal disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery Plus Chemothrapy (N=50)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 3 (3)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 9 (11)
Hemoglobin (Blood and lymphatic system disorders) | 47 (176)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 34 (62)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 45 (101)
Platelets (Blood and lymphatic system disorders) | 33 (109)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Vasovagal episode (Cardiac disorders) | 1 (1)
Cardiac left ventricular function (Cardiac disorders) | 1 (1)
Edema (Cardiac disorders) | 6 (6)
Hypertension (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Peripheral arterial ischemia (Cardiac disorders) | 1 (1)
Thrombosis/embolism (Cardiac disorders) | 4 (4)
Prothrombin time (PT) (Blood and lymphatic system disorders) | 1 (1)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 44 (111)
Fever (General disorders) | 12 (13) — (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L)
Rigors, chills (General disorders) | 1 (1)
Sweating (diaphoresis) (General disorders) | 3 (4)
Weight loss (General disorders) | 11 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 34 (37)
Bruising (in absence of grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 2 (2)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3 (6)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 8 (9)
Hot flashes/flushes (Endocrine disorders) | 4 (6)
Anorexia (Gastrointestinal disorders) | 33 (56)
Constipation (Gastrointestinal disorders) | 28 (45)
Dehydration (Gastrointestinal disorders) | 6 (8)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 28 (56)
Dyspepsia/heartburn (Gastrointestinal disorders) | 8 (9)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 4 (7)
Flatulence (Gastrointestinal disorders) | 3 (3)
Ileus (or neuroconstipation) (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 42 (91)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 30 (61)
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 10 (16)
Vomiting (Gastrointestinal disorders) | 30 (54)
Hematuria (in the absence of vaginal bleeding) (Blood and lymphatic system disorders) | 2 (2)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Vaginal bleeding (Blood and lymphatic system disorders) | 2 (2)
Alkaline phosphatase (Hepatobiliary disorders) | 13 (22)
Bilirubin (Hepatobiliary disorders) | 4 (4)
Hypoalbuminemia (Hepatobiliary disorders) | 25 (55)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 26 (58)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 23 (52)
Catheter-related infection (Infections and infestations) | 1 (1)
Febrile neutropenia (Infections and infestations) | 3 (3) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Infection (Infections and infestations) | 2 (2) — (documented clinically or microbiologically) with grade 3 or 4 neutropenia (ANC <1.0 x 10e9/L)
Infection without neutropenia (Infections and infestations) | 16 (29)
Infection/Febrile Neutropenia-Other (Specify, vag. yeast infection) (Infections and infestations) | 3 (4) — "Thrush", zoster, herpes L butt
Hypercalcemia (Metabolism and nutrition disorders) | 1 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 23 (44)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (15)
Hyponatremia (Metabolism and nutrition disorders) | 17 (22)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 9 (10)
Musculoskeletal-Other (Specify, fracture of L. fibula) (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (incoordination) (Nervous system disorders) | 4 (4)
Confusion (Nervous system disorders) | 5 (5)
Dizziness/lightheadedness (Nervous system disorders) | 7 (9)
Insomnia (Nervous system disorders) | 6 (8)
Mood alteration-anxiety, agitation (Nervous system disorders) | 2 (2)
Mood alteration-depression (Nervous system disorders) | 3 (5)
Neurology-Other (Specify, largyngitis, voice hoarseness; neurology: Tinnitus L>R ) (Nervous system disorders) | 2 (2)
Neuropathy - motor (Nervous system disorders) | 2 (2)
Neuropathy-sensory (Nervous system disorders) | 29 (48)
Cataract (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Tearing (watery eyes) (Eye disorders) | 2 (2)
Vision-blurred vision (Eye disorders) | 4 (4)
Vision-flashing lights/floaters (Eye disorders) | 1 (1)
Abdominal pain or cramping (Gastrointestinal disorders) | 19 (29)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 33 (93)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Chest pain (non-cardiac and non-pleuritic) (General disorders) | 2 (2)
Earache (otalgia) (Ear and labyrinth disorders) | 1 (1)
Headache (Nervous system disorders) | 9 (12)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 11 (18)
Pain-Other (Specify, Back Pain; Neck; Flank R; Pain in right rib ) (General disorders) | 4 (4)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rectal or perirectal pain (proctalgia) (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice changes/stridor/larynx (e.g., hoarseness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 3 (4)
Urinary retention (Renal and urinary disorders) | 5 (5)
Vaginitis (not due to infection) (Reproductive system and breast disorders) | 1 (1)
Sexual/Reproductive Function-Other (Specify, Amenorrhea) (Reproductive system and breast disorders) | 1 (1)
Dermatology/Skin-Other (Specify, Head Rash; pain: port problems, pain, redness ) (Skin and subcutaneous tissue disorders) | 2 (2)
Gastrointestinal-Other (Specify, dental extraction; early satiety; bloating) (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No